CLINICAL TRIAL: NCT02690389
Title: The Sedation Effect of Electro-acupuncture on Bilateral Zusanli (ST 36) and Neiguan (PC 6) in General Anesthesia May Not be Mediated by the Benzodiazepines- GABA Pathway
Brief Title: Electro-acupuncture and Flumazenil's Effect on Sedation
Acronym: EA&FLUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Yin Liu (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. Yin Liu, Associate Professor, Chief of Clinical Research, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SiChuanCHRI001
Record Dates: First submitted 2016-01-28; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Acupuncture; General Anaesthesia; Sedation
Keywords: Acupuncture; Flumazenil; Narcotrend; General Anaesthesia; Sedation
MeSH Terms: interventions — Flumazenil; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): standard procedure is used
- Flumazenil only group (Sham Comparator): flumazenil is given
  Interventions: Drug: Flumazenil
- control with acupuncture (Active Comparator): control with acupuncture
  Interventions: Procedure: Acupuncture
- control with acupuncture and flumazenil (Active Comparator): control with acupuncture and flumazenil
  Interventions: Drug: Flumazenil; Procedure: Acupuncture

INTERVENTIONS:
Drug: Flumazenil — used alone or with acupuncture
  Arms: Flumazenil only group; control with acupuncture and flumazenil
Procedure: Acupuncture — used alone or with flumazenil
  Arms: control with acupuncture; control with acupuncture and flumazenil

SUMMARY:
Object: To explore the mechanism of the electro-acupuncture (EA) induced sedation effect in general anaesthesia through investigating the role of the Benzodiazepines-GABA system.

Method: 80 patients undergoing abdominal surgery were randomly divided into four groups (n=20): C group (propofol only group), F group (propofol + flumazenil group), EA group (propofol + electro-acupuncture group), and EA+F group (propofol + electro-acupuncture + flumazenil group). Before induction, acupuncture needles were inserted at the points of Zusanli (ST 36) and Neiguan (PC 6) bilaterally to elicit"DeQi". Target-controlled infusion (TCI) of propofol was used for the induction and maintenance of anaesthesia. After 15minutes, equilibrium of Narcotrend Index (NT index) was achieved, patients were then assigned to receive different interventions. In EA group and EA+F group, patients received EA for 30 minutes under general anaesthesia, and flumazenil with the dosage of 0.1mg/kg was added in the latter at the end of EA. In C group and F group, patients didn't receive EA, and flumazenil with the dosage of 0.1mg/kg was administered in F Group at the same time point with EA+F group. HR, MAP and NT index were recorded at different time points up to 30 minutes after the end of EA.

ELIGIBILITY:
Inclusion Criteria:

* 80 abdominal surgical patients
* aged 30 to 60 years old,
* weighing 50-70Kg,
* ASA I-Ⅱ, who scheduled to receive general anaesthesia were enrolled to this trial.

Exclusion Criteria:

* Hypertension or severe heart and lung diseases,
* Conditions that might affect the consciousness or NT index, such as seizures, psychosis, brain lesions, and treatment with sedative drugs,
* Contraindications to acupuncture, such as severe hemorrhagic disease, hyper-sensitive patient, and tumor or ulcer exist on the skin of the acupuncture points.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
depth of general anaesthesia | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: yin liu, PhD, Principal Investigator — Sichuan University
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Data will not be share until it is published